CLINICAL TRIAL: NCT01722812
Title: An Exploratory Study Evaluating the Efficacy of Cromoglicate Cream Compared to Cream Vehicle in the Treatment of Itch in Psoriasis
Brief Title: Cromoglicate in Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0075-34
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2022-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Cromolyn Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (left) / Cromoglicate (right) (Other): Placebo (on a lesion on left body side), Cromoglicate (on a lesion on right body side)
  Interventions: Drug: Placebo
- Placebo (right) / Cromoglicate (left) (Other): Placebo (on a lesion on right body side), Cromoglicate (on a lesion on left body side)
  Interventions: Drug: Cromoglicate

INTERVENTIONS:
Drug: Cromoglicate — Twice daily topical treatment for 14 days
  Arms: Placebo (right) / Cromoglicate (left)
Drug: Placebo — Twice daily topical treatment for 14 days
  Arms: Placebo (left) / Cromoglicate (right)

SUMMARY:
The purpose of this exploratory study is to investigate the clinical efficacy of cromoglicate cream compared to cream vehicle in the treatment of itch in psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent has been obtained
* Age 18 years or above
* Either sex
* Any race or ethnicity
* Attending hospital outpatient clinic or the private practice of a dermatologist
* Clinical diagnosis of stable plaque psoriasis of at least 6 months with a symmetric distribution
* Two treatment areas with a symmetrical distribution each corresponding to 2-3% BSA (Body Surface Area) and each including at least one itchy psoriasis plaque
* Itchy psoriasis on both intended treatment areas of at least 40mm on the Visual Analogue Scale (VAS) with a maximum difference of 10mm on the visual analogue scale between each of the two treatment areas
* Disease severity graded mild, moderate or severe according to the Physician's global assessment (PGA) of disease severity on psoriasis plaques on each of the two treatment areas. The disease severity must be the same for both treatment areas

Exclusion Criteria:

* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation:

  * etanercept - within 4 weeks prior to randomisation
  * adalimumab, infliximab - within 8 weeks prior to randomisation
  * ustekinumab - within 16 weeks prior to randomisation
  * other products - 4 weeks/5 half-lives (whichever is longer)
* Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, methotrexate, ciclosporin, fumaric acid derivatives, and other immunosuppressants) within 4 weeks prior to randomization
* Any topical treatment of the treatment areas (except for emollients) within 2 weeks prior to randomisation.
* Treatment with therapies, whether marketed or not, with a possible effect on itch within the following time periods prior to randomisation:

  * antihistamines - within 1 week prior to randomisation
  * gabapentin - within 4 weeks prior to randomisation
* Subjects who have received treatment with any non-marketed drug substance (i.e. a drug which has not yet been made available for clinical use following registration) within the 4-week period prior to randomisation or longer, if the class of substance required a longer treatment free period as defined in exclusion criterion 1 for biological treatments
* PUVA (Psoralen and Ultraviolet A Radiation) or Grenz ray therapy within 4 weeks prior to randomisation.
* UVB therapy within 2 weeks prior to randomisation
* Planned initiation of, or changes to concomitant medication that could affect psoriasis vulgaris (e.g., beta blockers, ACE inhibitors, anti-malaria drugs, lithium) within 2 weeks prior to randomisation
* Subjects with current participation in any other interventional clinical trial
* Subjects with any of the following conditions present on the treatment areas: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, icthyosis, ulcers and wounds
* Other inflammatory skin disorders (e.g. seborrhoeic dermatitis or contact dermatitis) on the treatment area that may confound the evaluation of psoriasis
* Subjects with a history of serious allergy, allergic skin rash or sensitivity to any component of the investigational products or formulations being tested
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Current diagnosis of erythrodermic, exfoliative, guttate or pustular psoriasis
* Planned exposure to the sun during the study that may affect psoriasis vulgaris (i.e., normal lifestyle outdoor activities are permitted but deliberate exposure to sunlight or artificial ultraviolet light should be avoided)
* Subjects previously randomised into this trial
* Not all of the exclusion criteria listed due to limited space

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in visual analogue scale | Baseline to week 2

SECONDARY OUTCOMES:
Evaluation of change in 4-point itch scale, 7-point itch scale, duration of itch and comparison of treated areas | Baseline to week 2

CONTACTS AND LOCATIONS:
Locations (1):
- Allergie-Centrum-Charité, Department of Dermatology and Allergy, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No